CLINICAL TRIAL: NCT00876681
Title: Ultrasound Guidance Versus Electrical Stimulation for Continuous Popliteal-Sciatic Nerve Blocks: A Randomized, Controlled Trial
Brief Title: Ultrasound Guidance Versus Electrical Stimulation for Continuous Popliteal-Sciatic Nerve Blocks
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Brian Ilfeld, M.D., M.S./ Principal Investigator, University of California, San Diego, Department of Anesthesiology
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Popliteal Catheter: US vs. NS
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2009-10-08 (Estimated); Status verified 2009-10

CONDITIONS: Postoperative Pain; Foot Numbness
Keywords: Catheter; Ultrasound-guidance; Nerve Stimulation; Electrical stimulation; nerve block; UCSD; Orthopedic surgery; Foot/ankle pain; Foot/ankle numbness; Popliteal-Sciatic Catheters
MeSH Terms: conditions — Pain, Postoperative | interventions — Electric Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1. Ultrasound (Active Comparator): Ultrasound method of placement is selected randomly, using a computer program. The patient is asked their pain and discomfort using a 0-10 scale where 0=no pain/discomfort and 10=worst pain/discomfort imaginable. The patient is asked this question prior to surgery, but after catheter placement and then again the first day after surgery. Time of placement is also measured and begins when the ultrasound probe first touches the skin. Patients are also asked the numbness of their foot and toes based on a 0-10 scale where 0=no numbness and 10=completely numb.
  Interventions: Procedure: Popliteal catheter placed via ultrasound or electrical stimulation
- 2. Electrical Stimulation (Active Comparator): Electrical stimulation (nerve stimulation) method of placement is selected randomly, using a computer program. The patient is asked their pain and discomfort using a 0-10 scale where 0=no pain/discomfort and 10=worst pain/discomfort imaginable. The patient is asked this question prior to surgery, but after catheter placement, and then again the first day after surgery. Time of placement is also measured and begins when the nerve stimulation needle first touches the skin. Patients are also asked the numbness of their foot and toes based on a 0-10 scale where 0=no numbness and 10=completely numb.
  Interventions: Procedure: Popliteal catheter placed via ultrasound or electrical stimulation

INTERVENTIONS:
Procedure: Popliteal catheter placed via ultrasound or electrical stimulation — Patients will be randomized to one of two groups: Popliteal-sciatic catheter placed via ultrasound-guidance or placed via electrical stimulation. All patients will be given 40ml of 1.5% mepivicaine prior to surgery and then given a pain pump after surgery containing 0.2% ropivacaine. The patients pain scores will be assessed just prior to surgery and the day following surgery. The time of catheter placement and numbness the patient is experiencing in their foot and toes is also assessed and recorded by research staff.

SUMMARY:
Research study to determine if pain relief following foot and/or ankle surgery is influenced by the technique used to place perineural catheter. The catheters are placed using ultrasound-guidance or nerve stimulation and the method is selected at random using a computer program. This may help to determine if one of these methods is associated with an increased success rate and incidence of foot numbness during the infusion.

DETAILED DESCRIPTION:
Specific Aim 1: To determine the relationship between perineural catheter placement technique (ultrasound-guidance and electrical stimulation) and quality of postoperative analgesia during continuous popliteal-sciatic nerve blocks following moderate-to-severely painful orthopedic surgery.

Hypothesis 1: When inserting a perineural catheter for a continuous peripheral nerve block, the use of electrical stimulation, as compared with ultrasound-guidance, is associated with decreased pain the morning following moderate-to-severely painful orthopedic surgery as measured with a numeric rating scale.

Specific Aim 2: To determine the relationship between perineural catheter placement technique (ultrasound-guidance and electrical stimulation) and degree of sensory deficit during continuous popliteal-sciatic nerve blocks following moderate-to-severely painful orthopedic surgery.

Hypothesis 2: When inserting a perineural catheter for a continuous peripheral nerve block, the use of electrical stimulation, as compared with ultrasound-guidance, is associated with increased sensory deficit the day following moderate-to-severely painful orthopedic surgery as measured with a simple 0-10 scale (0=no numbness; 10=completely insensate) of the part of the foot with the greatest sensory deficit at the time of the data-collection phone call.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing surgery with a planned popliteal-sciatic perineural catheter for postoperative analgesia
* Expected postoperative pain to be at least moderate in severity the day following surgery (often not adequately treatable with oral analgesics alone)
* Age 18 years or older

Exclusion Criteria:

* Pregnancy
* Inability to communicate wiht the investigators and hospital staff
* Incarceration
* Current chronic opioid use (daily opioid equivalent of >10mg oxycodone for more than the previous four weeks)
* History of alcohol or opioid abuse
* Neuropathy in the surgical extremity
* Any physical, mental or medical conditions which may confound quantifying postoperative pain resulting from surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
The primary outcome measurement will be the average pain in the three hours previous to a phone call the day following surgery as measured on a numeric rating scale (NRS, 0-10, 0=no pain, 10=worst imaginable pain). | 3 hours on day following surgery

SECONDARY OUTCOMES:
Sensory deficit in the operative limb the day following surgery as measured with a simple 0-10 scale (0=no numbness; 10=completely insensate) of the part of the foot with the greatest sensory deficit at time of the data collection phone call. | 1 day
Time for catheter placement. Time will begin when probe is placed on skin for the ultrasound-guidance method and when the nerve stimulation needle is placed on the skin for the electrical stimulation method. | 30 minutes
Catheter placement success rate as assessed by attending physician who will test for sensory deficit. | 30 minutes
Worst pain experienced since the surgery in the surgical limb as measured on the 0-10 NRS as assessed by the research staff when they call the patient the day following surgery. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Brian M Ilfeld, M.D., M.S., Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Medical Center, San Diego, California, United States

REFERENCES:
- [Derived] Mariano ER, Loland VJ, Sandhu NS, Bishop ML, Lee DK, Schwartz AK, Girard PJ, Ferguson EJ, Ilfeld BM. Comparative efficacy of ultrasound-guided and stimulating popliteal-sciatic perineural catheters for postoperative analgesia. Can J Anaesth. 2010 Oct;57(10):919-26. doi: 10.1007/s12630-010-9364-7. Epub 2010 Aug 11. PMID 20700680